CLINICAL TRIAL: NCT01736878
Title: Randomized Double-blind Placebo Controlled Phase II Study to Evaluate the Efficacy and Safety of Sorafenib Treatment in Patients With Advanced (Recurrent, Persistent and/or Metastasizing) Medullary Thyroid Carcinoma
Brief Title: Efficacy and Safety Study of Sorafenib to Treat Advanced Medullary Thyroid Carcinoma
Acronym: SUMMIT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to unanticipated hassle in patient recruitment.
Sponsor: Eanm Research Ltd (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EARL-2; 2011-006250-90 (EudraCT Number)
Record Dates: First submitted 2012-10-23; First posted 2012-11-29 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Medullary Thyroid Carcinoma
Keywords: Medullary Thyroid Carcinoma; Sorafenib; Efficacy
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib tablets (Experimental): Oral administration of Sorafenib tablets, 400 mg bid, until disease progression or unacceptable toxicity
  Interventions: Drug: Sorafenib
- Placebo tablets (Placebo Comparator): Oral administration of Placebo tablets until disease progression, afterwards continuation with Sorafenib at the discretion of the investigator
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib

SUMMARY:
The purpose of his study is to evaluate the efficacy and safety of Sorafenib versus placebo in subjects with locally advanced medullary thyroid cancer (MTC). The primary study objective is to compare the Progression-free Survival (PFS) of the Sorafenib treatment group with the placebo treatment group in patients with advanced MTC.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient ≥ 18 years of age
* Histologically confirmed medullary thyroid carcinoma
* Recurrent or persistent local disease and/or distant metastases
* No more than one prior line of systemic therapy
* Best available supportive care to control (endocrine) symptoms
* At least one defined lesion in CT or MRI evaluable for Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or at least one defined lesion in CT or MRI not evaluable by RECIST in combination with elevated tumour markers
* Progression within previous 12 months
* Hb > 8g/dl, white blood cells (WBC) >3.000 cells/mm³ (ANC > 1.500 cells/mm³), platelets > 100.000 cells/mm³, bilirubin < 2mg/dl, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN)
* Performance status: WHO ≤ 2; Karnofsky index ≥ 50%
* Sufficient renal function (creatinin <1.5 mg/dl and creatinin clearance > 30ml/min)
* International normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 x ULN
* No acute infections
* Staging studies (MRT or CT and Calcitonin or CEA) completed within four weeks of protocol randomisation
* Women of childbearing potential with negative serum pregnancy test
* Women and men of childbearing potential using adequate contraception
* Signed and dated written informed consent

Exclusion Criteria:

* Unresolved toxicity (i.e. neurotoxicity) attributed to any prior therapy higher than National Cancer Institute-Common Toxicity Criteria for Adverse Effects (NCI-CTCAE version 4) Grade 2 (excluding cases of alopecia)
* Patients with history of allergic or hypersensitivity reaction to study drug or placebo or their excipients
* Current participation in another investigational trial
* Patients with significant cardiovascular disease
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy other than beta-blockers or digoxin
* Congenital long corrected QT interval (QTc) syndrome, history of drug induced QTc prolongation, or QTc interval unmeasurable or more than 450 ms
* Abnormal serum electrolytes such as potassium, magnesium and calcium
* Uncontrolled hypertension, despite optimal management
* Major surgery, open biopsy, or significant traumatic injury within 30 days prior to randomization
* Non-healing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy disorder
* Hemorrhage/bleeding event ≥ Grade 3
* Thrombotic or embolic events including transient ischemic attacks within the past 6 months
* Subjects with symptomatic brain metastases or Subjects with brain metastases under corticosteroid treatment
* Pregnant or breast-feeding patients
* Patients with uncontrolled infections
* Known HIV infection or infection with hepatitis B or C
* Immunosuppression
* Subjects with seizure disorder requiring medication • Subjects undergoing renal dialysis
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Any malabsorption condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | from the date of randomisation until the date of radiological or biochemical progression or death. An average of 9 months is assumed.
  The proportion of patients with PFS in the Sorafenib group and the Placebo group will be compared by log rank test and Kaplan-Meier plot.

SECONDARY OUTCOMES:
Time to Progression (TPP) | from the date of randomisation until the date of confirmed radiological or biochemical progression. An average of 9 months is assumed.
  The average TTP in the Sorafenib group and the Placebo group will be compared.

OTHER OUTCOMES:
Overall Survival (OS) | from the date of randomisation until the date of death due to any cause. Final assessment at the end of study after approximately 36 months.
  The proportion of surviving patients in the Sorafenib group and the Placebo group will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ulm, Clinic for Nuclear Medicine, Ulm, Baden-Wurttemberg, Germany